CLINICAL TRIAL: NCT04365348
Title: Exploring the Psychological Impact of the COVID-19 Outbreak on COVID-19 Survivors and Their Families
Brief Title: The Psychological Impact of COVID-19 Outbreak on COVID-19 Survivors and Their Families
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant Professor, The University of Hong Kong
Other Study IDs: UW20-300
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Mental Health Wellness 1
Keywords: Stress; Anxiety; Depression; Families
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with COVID-19 diagnoses are treated under isolation in hospitals and with high-stress level. Currently, there is little information on the mental health implications of exposure amongst COVID-19 survivors and their family members. Research exploring the psychological impact amongst survivors of exposure to COVID-19 is desperately needed to understand the effects, mental health toll, and support required in survivors of COVID-19. This study aims to assess the psychological impact of the COVID-19 outbreak on COVID-19 survivors and their family members.

DETAILED DESCRIPTION:
Since the 2019 coronavirus disease (COVID-19) was first reported, it has been rapidly transmitted and has aroused enormous global attention. Infected patients may develop severe and even fatal respiratory symptoms such as acute respiratory distress syndrome (ARDS) and acute respiratory failure, ending up in intensive care. Patients with COVID-19 diagnoses are treated under isolation in hospitals and with high-stress level. The stress and psychological impact on patients were also correlated significantly with several adverse psychological effects, such as fatigue, fear of social contact, poor sleep, loneliness, and depressed mood. The psychological impact of COVID-19 may also evolve and last for a prolonged period after discharge from the hospital. However, there is currently little information on the mental health implications of exposure amongst COVID-19 survivors and their family members. Research exploring the psychological impact amongst survivors of exposure to COVID-19 is desperately needed to understand the effects, mental health toll, and support required in survivors of COVID-19. This study aims to assess the psychological impact of the COVID-19 outbreak on COVID-19 survivors and their family members.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 survivors (i.e., diagnosed with COVID-19 and discharged from the hospital) and/or a family member of a COVID-19 survivor;
* Aged 18 years or above;
* No medical diagnosis of psychiatric illness

Exclusion Criteria:

• Refusal to give consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 Survivors: 300; Family members of COVID-19 Survivors:300
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Stress level | 1 month
  measured by the 10-item Perceived Stress Scale

SECONDARY OUTCOMES:
Stress level | 3 months
  measured by the 10-item Perceived Stress Scale
Negative emotion | 3 months
  measured by the 13-item Hospital Anxiety and Depression Scale
Psychological response to trauma | 1 month and 3 months
  measured by the 22-item Impact of Event Scale -Revised
Severity of insomnia symptoms and the associated daytime impairment | 1 month and 3 months
  measured by the 7-item Insomnia Severity Index
Resilience | 1 month and 3 months
  measured by the 2-item Connor-Davidson Resilience Scale
Quality of family functioning | 1 month and 3 months
  measured by 3-item Family Functioning Subscale
Social support | 1 month and 3 months
  measured by 6-item social support questionnaire
Psychological effects | 1 month and 3 months
  measured by 10-item outcome-based questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Agnes, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
It has not been mentioned in the participants' consent

REFERENCES:
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Chua SE, Cheung V, McAlonan GM, Cheung C, Wong JW, Cheung EP, Chan MT, Wong TK, Choy KM, Chu CM, Lee PW, Tsang KW. Stress and psychological impact on SARS patients during the outbreak. Can J Psychiatry. 2004 Jun;49(6):385-90. doi: 10.1177/070674370404900607. PMID 15283533